CLINICAL TRIAL: NCT07038941
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial of Single and Multiple Doses of CG2001 in Chinese Adult Male Participants With Androgenetic Alopecia
Brief Title: Phase I Clinical Trial of CG2001 in Chinese Adult Male Participants With Androgenetic Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Dayspring Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG2001-C-1
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Male Pattern of Hair Loss, Androgenic Alopecia; Androgenetic Alopecia (AGA)
Keywords: minoxidil; finasteride
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm 1 (Experimental): 5% minoxidil and 0.025% finasteride, 1 gram Only once on Day 1
  Interventions: Drug: CG2001
- Arm 2 (Experimental): 5% minoxidil and 0.05% finasteride, 1 gram Once a day from Day 1 to Day 7
  Interventions: Drug: CG2001
- Arm 3 (Experimental): 5% minoxidil and 0.075% finasteride, 1 gram Once a day from Day 1 to Day 7
  Interventions: Drug: CG2001
- Arm 4 (Experimental): 5% minoxidil and 0.1% finasteride, 1 gram Once a day from Day 1 to Day 7
  Interventions: Drug: CG2001
- Arm 5 (Experimental): 5% minoxidil and 0.1% finasteride, 1 gram Once a day on Day 1, twice daily on Day 2 to Day 6, once a day on Day 7
  Interventions: Drug: CG2001
- Arm 6 (Placebo Comparator): Placebo foam, 1 gram Once a day from Day 1 to Day 7
  Interventions: Drug: Placebo foam
- Arm 7 (Placebo Comparator): Placebo foam, 1 gram Once a day on Day 1, twice daily on Day 2 to Day 6, once a day on Day 7
  Interventions: Drug: Placebo foam

INTERVENTIONS:
Drug: CG2001 — combination of minoxidil and finasteride
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5
Drug: Placebo foam — Placebo foam
  Arms: Arm 6; Arm 7

SUMMARY:
This study is testing CG2001, a new medicine that is applied as a light foam to the scalp and is being developed to treat male-pattern hair loss (androgenetic alopecia). The main goals are to find out:

1. Whether single and repeated daily doses of CG2001 are safe and well-tolerated
2. How much of the drug, if any, enters the bloodstream (pharmacokinetics)

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included:

1. Voluntarily sign the informed consent form approved by the ethics committee before any research procedures begin;
2. Be able to understand and comply with the requirements of the protocol, and agree to cooperate in completing all research procedures for research visits;
3. Male, aged 18-65 years (including critical values);
4. Body mass index is 18-28 kg/m2 (including critical values), and weight must not be less than 50 kg;
5. Diagnosed with androgenic alopecia in accordance with the "Guidelines for the Diagnosis and Treatment of Androgenic Alopecia in Chinese" (2019), and manifested as frontal hairline recession or hair loss in the top scalp area, and meet the standards of grade III top type, grade IV and grade V of the Hamilton-Norwood classification;
6. Agree to use appropriate medical contraceptive methods to avoid pregnancy in female partners from the signing of the informed consent form until 28 days after the last dose.

Exclusion Criteria:

Participants who meet any of the following conditions are not eligible to participate in this study:

1. Allergic to minoxidil, finasteride or any component of the excipients, or allergic constitution;
2. Participants with any of the following conditions regarding past medical history, current medical history and treatment history of the skin (including the head skin) are not eligible to participate in this study; A. Participants who the investigator believes have scalp skin abnormalities or a history of scalp skin diseases that may interfere with the study evaluation; B. Participants with secondary alopecia such as malnutrition, drugs, endocrine (hypothyroidism or hyperthyroidism, hypoparathyroidism or hypopituitarism), iron deficiency anemia and systemic lupus erythematosus causing alopecia; C. Participants with alopecia areata, scarring alopecia or trichotillomania; D. Participants who have undergone hair transplantation, hair extensions, or need to wear a wig for a long time during the study treatment; E. Participants who have used systemic or topical corticosteroids or synthetic steroids for scalp within 3 months before screening; F. Participants who have received scalp radiation, phototherapy/laser, local injection of autologous platelet-rich plasma (PRP) or surgical treatment within 6 months before screening;
3. For other systemic past medical history, current medical history and treatment history, those with any of the following conditions cannot participate in this study:

   A. Underwent major surgery 2 months before screening, or lost blood or donated blood > 500mL within 3 months before the first dose; B. Had a history of drug abuse; C. Used any drug that inhibits or induces liver drug metabolizing enzymes within 14 days before the first medication, or used any drug that inhibits or induces liver drug metabolizing enzymes and the last medication time was less than 5 half-lives of the drug, whichever is the longest; D. Used any prescription drugs, over-the-counter drugs, Chinese patent medicines, any herbal products and health products within 14 days before the first medication; E. Has a history of varicocele, sexual dysfunction or infertility; F. Participant with severe respiratory, digestive, urinary, immune, blood, endocrine, metabolic, neurological and psychiatric diseases in the past or currently, or poor disease control, which the investigators assess will significantly affect the safety and/or compliance of the participants in participating in this study; G. Participant with a history of malignant tumors but clinically cured for 5 years, or participant with completely resected carcinoma in situ, localized prostate cancer that has received radical treatment and has no disease recurrence, and completely resected basal cell or squamous cell skin cancer can participate in this study;
4. Regarding laboratory examinations, participant who meet any of the following criteria are excluded; A. Complete blood count: hemoglobin <9 g/dL, platelets <90×109/L, white blood cells <3.0×109/L; B. Liver function: alanine aminotransferase or aspartate aminotransferase or total bilirubin >2 times the upper limit of normal value; C. Renal function: eGFR <60 mL/min/1.73m2; or abnormal blood creatinine and determined by the investigators to be clinically significant.

   D. Infectious disease examination: participant with active hepatitis B (positive hepatitis B surface antigen and hepatitis B virus deoxyribonucleic acid HBV DNA ≥ upper limit of normal value), or positive hepatitis C virus antibody (HCV-Ab) and positive hepatitis C virus (HCV) RNA result, or positive Treponema pallidum antibody, or positive human immunodeficiency virus (HIV) antibody test result; E. 12-lead electrocardiogram examination: the average value of QT interval (QTcF) after QT interval correction using Fridericia formula, QTcF>450 ms; F. Any result of breath alcohol test and urine drug screening is positive.
5. Participated in other interventional drug clinical trials and received the trial drugs within 3 months before the start of the trial;
6. Difficulty in venous blood collection (such as needle phobia, blood phobia, etc.);
7. The researcher believes that there are any other reasons that make the participant unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | From baseline to 4 days post last administration
  Incidence and severity of adverse events, vital signs, physical examination, laboratory tests, electrocardiogram, etc.

SECONDARY OUTCOMES:
Single dose: Area under the plasma concentration versus time curve | Within 1 hour before and 24 hours after intervention administration
Single dose: Peak Plasma Concentration | Within 1 hour before and 24 hours after intervention administration
Single dose: Time to first peak drug concentration | Within 1 hour before and 24 hours after intervention administration
Single dose: Terminal elimination half-life | Within 1 hour before and 24 hours after intervention administration
Single dose: Volume of Distribution | Within 1 hour before and 24 hours after intervention administration
Single dose: Clearance rate | Within 1 hour before and 24 hours after intervention administration
Single dose: Elimination rate | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Area under the plasma drug concentration versus time curve at steady state | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Peak Plasma Concentration; | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Trough Plasma Concentration | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Accumulation index | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Average steady-state plasma drug concentration | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Apparent volume of distribution at steady state | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Apparent clearance rate at steady state | Within 1 hour before and 24 hours after intervention administration
Multiple dose: Half-life at steady state | Within 1 hour before and 24 hours after intervention administration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Fang, MD, PhD, Principal Investigator — Peking University People's Hospital; Jianzhong Zhang, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China